CLINICAL TRIAL: NCT05822115
Title: Reduction of Breast Hypertrophy by Means of Coelioscopique Surgery
Acronym: R-HTM-R
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Groupe Hospitalier Nord-Essonne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-A01278-35
Record Dates: First submitted 2023-03-21; First posted 2023-04-20 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-03

CONDITIONS: Breast Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treated group (Experimental): Breast reduction
  Interventions: Device: Reduction of breast hypertrophy by means of laparoscopic

INTERVENTIONS:
Device: Reduction of breast hypertrophy by means of laparoscopic — The research procedure is a breast reduction performed by means of laparoscopic surgery.
  The project consists of removing a disc from the breast at the level of the base, thus causing peripheral skin slackening of 2 to 3 cm but circular. Both breasts are usually operated on at the same time. In case of asymmetry, only one side will be treated.
  Other Names: R-HTM-R

SUMMARY:
The objective of this interventional study is based on the hypothesis that coelioscopique surgery could be used to reduce breast hypertrophy.

This study can be expected to scientifically validate the use of laparoscopic surgery to obtain a clinical result in the context of reduction of medium volume breast hypertrophy.

DETAILED DESCRIPTION:
Breast reductions are common procedures. One of the main difficulties related to this surgery remains the healing, wide at the peri-areolar level, vertical at the sub-areolar level and in the sub-mammary fold. In addition, this intervention remains subject to the vagaries of hypertrophic or even keloidal healing, especially in young subjects.

On This study can be expected to scientifically validate the use of laparoscopic surgery to obtain a clinical result without scarring in the context of the reduction of medium volume breast hypertrophy.

Ultimately, the results of this study may serve as a basis for further research by proposing:

* Prophylactic mastectomies and immediate breast reconstruction without lateral scar and with a less visible sub-breast scar.
* A breast reduction in young patients before the skin undergoes the effects of the heaviness of the breasts.

ELIGIBILITY:
Inclusion criteria :

* Women over the age of 18.
* Category 1 or 2 according to the Regnault classification.
* C cup breast size or larger.
* Areola "looks ahead" i.e. a distance between point A (at the top of the areola) at the median suprasternal point of approximately 16 cm to 24 cm.
* Ptosis (distance between the lowest part of the breast and the submammary fold) of a maximum of 7cm (measured in a seated position).
* Expected correction of half ptosis with decrease of 1 to 3 cup sizes.
* Patient has good quality thick skin.
* Social security scheme.
* Patient requesting breast reduction.
* Patient having signed the free and informed consent.

Non inclusion criteria :

* Areola "look down"; point A more than 25 cm.
* Ptosis greater than or equal to 8 cm.
* Thin skin.
* Smoker.
* Patient under effects of anti-coagulant.
* Patient participating in another clinical study.
* Protected patient: adults under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision.
* Pregnant, lactating woman.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Photography of the scar | at 3 months
  centimeter

SECONDARY OUTCOMES:
Scar assessment | at 3 weeks
  number of scars
Resection weight | at 0 day
  Resection weight
Photography of Areola | at 3 weeks, 3 months and 1 year
  Centimeter
Scar lenght | at 3 weeks, 3 months and 1 year
  Centimeter
Blood loss | at 1 day
  the haemoglobin (hb) level
Pain scale | at 3 weeks, 3 months and 1 year
  0 (no pain) to 10 (very intense pain)
Satisfaction scale | at 3 weeks, 3 months and 1 year
  0 (dissatisfied) to 10 (satisfied)
Cancer | at day 0
  presence or absence
Macroeconomic impact | at 1 year
  length of hospital stay, duration of surgery
Scar thickness | at 3 weeks, 3 months and 1 year
  Centimeter

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Eric DUNET, Longjumeau, France

IPD SHARING:
Plan to Share IPD: No